CLINICAL TRIAL: NCT04470999
Title: Cellular Immune Profile Changes in Individuals With Active or Past COVID-19 Infection
Brief Title: Changes in Cellular Immune Profile During COVID-19 Infection
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to the move of clinical trial site. It will be resumed when the move is complete.
Sponsor: Serhat Gumrukcu, MD PhD (Other)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Sponsor-Investigator, Serhat Gumrukcu, MD PhD, Sponsor-Investigator, Seraph Research Institute
Organization: Seraph Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SRPH-CVD-01
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Covid19; SARS-CoV-2
Keywords: SARS-CoV-2; COVID; COVID19; Coronavirus; Cell therapy; Immunotherapy
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Venous blood and apheresis collection will be conducted
  Interventions: Other: Leukapheresis

INTERVENTIONS:
Other: Leukapheresis — Blood collection and PBMC collection via apheresis machine will be conducted
  Other Names: Mononuclear cell collection

SUMMARY:
Clinical specimens are collected from individuals either recovered from or with active SARS-CoV-2 infection to support process and analytical development for a potential cell-based immunotherapy in preclinical research, SRPH-CVD-01.

SRPH-CVD-01 is an allogeneic cell-based immunotherapy candidate to be investigated in a subsequent clinical trial under a future FDA IND to treat people suffering from COVID-19.

Enrolled participants provide a venous blood specimen (up to 40mL) to be used in preclinical studies and research and development of SRPH-CVD-01. Subjects may eventually be asked to undergo leukapheresis for peripheral blood mononuclear cell (PBMC) collection and their specimens will be used to further develop the SRPH-CVD-01 cell product, including a cGMP compliant process to be applied under the future FDA IND.

DETAILED DESCRIPTION:
This protocol is to collect blood and PBMC specimens from individuals with active of past COVID-19 infection. The first blood draw will be done at the first study visit and if eligible, the second collection will be done via leukapheresis at the second visit. The leukapheresis procedures will follow the facility's standard operating procedures and protocol requirements for leukapheresis.

Donors will be males or females between and including the ages of 18 years and 60 years. Volunteers will provide written informed consent and meet all inclusion and exclusion criteria. Each participant can be in the study for up to 180 days (6 months).

The study will be conducted in accordance with human research for the purposes of obtaining clinical specimens for research. There is no endpoint for this study, however, data collected from this study will include, but not be limited to, gender, demographics, medical history, clinical laboratory values, and volume of the blood collected. The data will be summarized in future studies reporting results from a future clinical trial under FDA IND.

ELIGIBILITY:
Inclusion Criteria:

* Male of female aged 18-60
* Documented current or past (max 3 months prior) diagnosis of COVID19
* Participants who has not participated in a cell or gene therapy trial for COVID19

Exclusion Criteria:

* Uncontrolled SARS symptoms
* Oxygen saturation (Pulse Ox) < 90%
* Uncontrolled diabetes
* Uncontrolled hypertension
* Active DIC, bleeding or coagulopathy which cannot be corrected with minimal intervention
* Symptomatic, uncontrolled or severe intercurrent illness that would compromise the ability to tolerate blood collection or leukapheresis procedure
* Systemic chemotherapy less than or equal to 2 weeks (6 weeks for clofarabine or nitrosoureas) or radiation therapy less than or equal to 3 weeks prior to leukapheresis
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test at screening
* Any patient that in the opinion of the investigator is not medically stable to undergo the leukapheresis procedure or will not comply with the visit schedules or procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cellular immune system profiling | Up to 20 days
  After the initial venous blood draw, the blood samples will be tested to measure the absolute count and percentage of B cells, monocytes, CD4+ and CD8+ T cells, gammadelta T (gdT) cells, CD3+CD56+ natural killer T (NKT) cells, and natural killer (NK) cells in total PBMCs.
  Data will describe the range of each cell population across participants.

SECONDARY OUTCOMES:
Innate immune system profiling | Up to 100 days
  Innate immune system cells (gdT, NKT, and NK) will be assessed for their SARS-CoV-2 antiviral activity by stimulation and immunophenotyping.
  Data will report the antiviral phenotypic characteristics of these cells.
Expansion of virus-specific innate immune cells | Up to 100 days
  Virus-specific innate immune cells that are relevant to SRPH-CVD-01 clinical product candidate will be expanded under various conditions to assess their therapeutic and protective potential against COVID-19. Data will report the expansion rate of SRPH-CVD-01 cells.
  These cell will also help validate the assays and processes for the development of the SRPH-CVD-01 cell product to be used in a future clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Gumrukcu, MD PhD, Principal Investigator — Seraph Research Institute
Locations (1):
- Seraph Research Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No